CLINICAL TRIAL: NCT00595439
Title: The Association Between Focal Dystonia (FD) and Complex Regional Pain Syndrome (CRPS)
Brief Title: Association Between Focal Dystonia and Complex Regional Pain Syndrome
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080040; 08-N-0040
Record Dates: First submitted 2007-12-28; First posted 2008-01-16 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-10-05

CONDITIONS: Focal Dystonia; Peripheral Nervous System Disease
Keywords: Sensory Evoked Potentials (SEPs); Electromyogram; Transcranial Magnetic Stimulation (TMS); Complex Regional Pain Syndrome; Focal Hand Dystonia; Focal Dystonia; Chronic Regional Pain Syndrome; CRPS
MeSH Terms: conditions — Dystonic Disorders; Peripheral Nervous System Diseases; Complex Regional Pain Syndromes; Dystonia, Focal, Task-Specific

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will investigate differences among people with focal dystonia (FD), complex regional pain syndrome (CRPS) and people who have both conditions to learn more about the cause of both disorders.

Participants undergo the following procedures in five visits:

* Electroencephalography (EEG). Electrodes (metal discs) are placed on the scalp with an electrode cap, a paste or a glue-like substance. The spaces between the electrodes and the scalp are filled with a gel that conducts electrical activity. Brain waves are recorded while the subject lies quietly and sensory stimulation is applied to the thumb or finger.
* Magnetic resonance imaging (MRI). This test uses a magnetic field and radio waves to obtain images of body tissues and organs. The patient lies on a table that can slide in and out of the scanner, wearing earplugs to muffle loud knocking and thumping sounds that occur during the scanning process. The procedure lasts about 45 minutes, during which time the patient will be asked to lie still for up to 15 minutes at a time.
* Transcranial magnetic stimulation (TMS). An insulated wire coil is placed on the scalp and a brief electrical current is passed through the coil. The current induces a magnetic field that stimulates the brain. There may be a pulling sensation on the skin under the coil and a twitch in muscles of the face, arm or leg. During the stimulation, subjects may be asked to keep their hands relaxed or to contract certain muscles.
* Peripheral electrical stimulation. In two experiments, TMS is combined with peripheral electrical stimulation, similar to what is used in nerve conduction studies, to the median nerve at the wrist. There may be muscle twitching.
* Surface electromyography. For TMS tests and peripheral electrical stimulation, electrodes are filled with a conductive gel and taped to the skin to record the electrical activity of three muscles on the right hand.
* Needle EMG. A needle is inserted into a muscle to record the electrical activity.
* Nerve conduction studies. A probe is placed on the skin to deliver a small electrical stimulus, and wires are taped to the skin record the nerve impulses. These studies measure the speed with which nerves conduct electrical impulses and the strength of the connection between the nerve and the muscles.
* Skin biopsy. Two sites are biopsied. A local anesthetic is given to numb the area and a 1/4-inch piece of skin is removed with a special tool.
* JVP domes. Subjects are tested for their ability to discriminate sensory stimuli in the affected region and on the other side of it. They are asked to discriminate between stamps with grooves of different widths that are applied to the hands or feet.

DETAILED DESCRIPTION:
OBJECTIVE

Dystonia is generally regarded as a motor execution abnormality due to a central nervous system dysfunction in the cortico-striato-thalamo-cortical motor loop. Regional traumas are considered to be risk factors for the development of focal dystonia (FD) in the affected limb. Since focal limb traumas are also associated with complex regional pain syndrome (CRPS), there may be a common underlying pathology in both conditions. In CRPS, many patients have a small fiber neuropathy. The goal of the proposed research is to distinguish (discriminate) among the three disease categories (FD, FD+CRPS, CRPS), to find out whether FD and CRPS share a common physiological substrate and represent two sides of a spectrum, and to see which clinical situations may be secondary to an underlying small fiber neuropathy. Independent studies will be conducted in patients with affected upper limbs and in those with affected lower limbs.

STUDY POPULATION

We intend to perform two studies on overall 90 subjects. One study will assess the affected upper limb in 15 patients with unilateral focal dystonia, 15 patients with CRPS and 15 patients with focal dystonia and CRPS, while the second study will test the affected lower limb in 15 patients with unilateral focal dystonia, 15 patients with CRPS and 15 patients with focal dystonia and CRPS in the lower limb.

DESIGN

We propose to explore the central aspects (somatosensory evoked potentials, SEPS, and transcranial magnetic stimulation, TMS) in patients with upper limb disorders, because the cortical representation of hand muscles is easier to study than the lower limb muscle representations. In contrast, the peripheral studies (quantitative EMG and nerve conduction) will be performed in patients with lower limb disorders, due to length, accessibility and separation of pure motor and sensory nerves in the leg.

OUTCOME MEASURES

The primary outcome measure for the central nervous system features (the upper limb assessment) will be the difference in EEG dipole localization of the SEPs from thumb and index finger between the three groups to assess possible disturbances of cortical representation in the primary sensory cortex. TMS measures will be exploratory.

The primary outcome measure of the lower limb testing will be the duration of motor unit action potentials (MUAP) to assess differences and subtle lesions, which were not picked up in clinical routine due to bigger confidence intervals of the single parameter.

The unaffected side is the primary target of this study since we are looking for an underlying substrate; however, all clinical tests will be performed bilaterally (if tolerated by the subjects) and the comparison of both sides will be a secondary outcome measure.

ELIGIBILITY:
* INCLUSION CRITERIA:

PATIENTS WITH FOCAL DYSTONIA (ONLY):

* Age 18 years or older
* Presence of FD and no CRPS

PATIENTS WITH CRPS (ONLY):

* Age 18 years or older
* Presence of CRPS and no FD

PATIENTS WITH DYSTONIA AND CRPS (CRPS + DYSTONIA):

* Age 18 years or older
* Presence of FD and CRPS in the same limb

EXCLUSION CRITERIA:

* Concurrent significant medical, surgical, neurologic or psychiatric condition
* Taking the following medications: anxiolytics, antipsychotics, antiparkinson, hypnotics, stimulants, and/or antihistamines
* Taking antidepressants or anticonvulsants needs to be discussed specifically in each patient
* Received botulinum toxin injection within 3 months of starting the protocol
* For TMS: Presence of pacemaker, implanted medical pump, metal plate or metal object in skull or eye
* History of seizure disorder
* No known history of hearing loss
* For MRI: Presence of pacemakers or other implanted electrical devices, brain stimulators, dental implants, aneurysm clips, metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pumps, or shrapnel fragments. Welders and metal workers are also at risk for injury because of possible small metal fragments in the eye of which they may be unaware.
* Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2007-12-21; Primary Completion 2009-10-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hallett M. Dystonia: abnormal movements result from loss of inhibition. Adv Neurol. 2004;94:1-9. No abstract available. PMID 14509648
- [Background] Bressman SB. Dystonia genotypes, phenotypes, and classification. Adv Neurol. 2004;94:101-7. No abstract available. PMID 14509661
- [Background] Rothwell JC, Obeso JA, Day BL, Marsden CD. Pathophysiology of dystonias. Adv Neurol. 1983;39:851-63. No abstract available. PMID 6660125